CLINICAL TRIAL: NCT00397410
Title: Compliance With and Effect of Soft and Hard Hip Protectors in Norwegian Nursing Homes
Brief Title: Prevention of Hip Fractures With Soft and Hard Hip Protectors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Oslo University College (Other)
Responsible Party: Principal Investigator, Hege Bentzen, PhDcandidate, Norwegian Institute of Public Health
Allocation: Randomized | Masking: None
Other Study IDs: 2004-2-0284
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Hip Fractures; Prevention
Keywords: hip protectors; uptake and adherence; Nursing home residents; efficacy; prevention
MeSH Terms: conditions — Hip Fractures

INTERVENTIONS:
Device: Hip protectors

SUMMARY:
The aim of this study is to compliance with and effect of soft and hard hip protectors in Norwegian nursing homes.

DETAILED DESCRIPTION:
Hip fractures are a major cause of disability and functional limitation. Hip protectors have shown to have the potential to lower the risk of a fracture by reducing the impact on the hip region during falls, but low uptake and adherence have been a problem.

Changing the hip protector's design might give a higher uptake and adherence. The aim of this study is to compare uptake, adherence and effect of soft and hard hip protectors in Norwegian nursing homes. Because a soft hip protector seems to be more comfortable, we expect a higher uptake and adherence with the soft hip protector, specially when it comes to 24 hour use. If the soft hip protector has the same protective quality as the hard hip protector, the soft hip protector will be a better alternative than the hard one.

This cluster randomized study is performed in 18 Norwegian nursing homes in 2 municipalities. The study started May 15. 2006 and will end November 30. 2006.

All permanent residents are invited to participate in the study either as a user of hip protector or as a non user.

ELIGIBILITY:
Inclusion Criteria:

* all permanent residents in the the participating nursing homes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1236 (Actual)
Dates: Start 2005-05; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Uptake and adherence with soft and hard hip protectors
Effect of soft and hard hip protectors in protected and unprotected falls

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Forsen, PHd, Principal Investigator — National Institute of public Health
Locations (1):
- Norwegian Institute of public Health, Oslo, Norway